CLINICAL TRIAL: NCT04460547
Title: Worldwide Trends on COVID-19 Research After the Declaration of COVID-19 Pandemic: An Observational Study
Brief Title: Worldwide Trends on COVID-19 Research After the Declaration of COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qassim University (Other)
Responsible Party: Principal Investigator, Dr Shiva Shankar Bugude, Assistant Professor, Qassim University
Other Study IDs: COAHS
Record Dates: First submitted 2020-07-03; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
Keywords: Research trends, COVID-19, Pandemic, Interventional studies, Observational studies
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; oplunofusp; Ivermectin; Interferon beta-1a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Completed Interventional studies: Interventional studies in the WHO-compliant registries database which are registered and completed before 11th March 2020.
  Interventions: Drug: Convalescent Plasma Transfusion; Drug: Hydroxychloroquine; Drug: DAS181; Drug: Ivermectin; Drug: Interferon Beta-1A
- Completed Observational studies: Observational studies in the WHO-compliant registries database which are registered and completed before 11th March 2020.
  Interventions: Drug: Convalescent Plasma Transfusion; Drug: Hydroxychloroquine; Drug: DAS181; Drug: Ivermectin; Drug: Interferon Beta-1A

INTERVENTIONS:
Drug: Convalescent Plasma Transfusion — Convalescent Plasma Transfusion to COVID-19 infected patients.
Drug: Hydroxychloroquine — Hydroxychloroquine administration to COVID-19 infected patients.
Drug: DAS181 — DAS181 administration to COVID-19 infected patients.
Drug: Ivermectin — Ivermectin administration to COVID-19 infected patients.
Drug: Interferon Beta-1A — Interferon Beta-1A administration to COVID-19 infected patients.

SUMMARY:
On 11th of March 2020, WHO characterized COVID-19 infection as a Pandemic. After the COVID-19 infection is declared as a Pandemic there was an outburst regarding COVID-19 Research. The Research interest led to registration of Interventional and Observational studies world wide. There are constant efforts by Health care workers to seek information regarding the Interventional and Observational studies which can help in decision making regarding effective handling of COVID-19 infected patients. It is also important to track on the happenings in various frontiers of COVID-19 Research in view of historical interest and clinical relevance. This Observational Cross sectional study aims to explore the completed Researches in WHO-compliant registries to understand the trends of COVID-19 Research. This study aims to get a birds eye view of ongoing COVID-19 Research scenario worldwide. This study results can directly benefit the worldwide Academicians and Health Care Professionals to understand the ongoing COVID-19 Research trends.

DETAILED DESCRIPTION:
On 11th of March 2020, WHO characterized COVID-19 infection as a Pandemic. After the COVID-19 infection is declared as a Pandemic there was an outburst regarding COVID-19 Research. The Research interest led to registration of Interventional and Observational studies world wide.

AIMs & Objectives of the Study This Observational Cross sectional study aims to explore the completed Researches in WHO-compliant registries to understand the trends of COVID-19 Research.

This study results can directly benefit the worldwide Academicians and Health Care Professionals to understand the ongoing COVID-19 Research trends.

Primary Outcomes of the Study To understand the geographical distribution of the interventional studies after 11th of March 2020.

To understand the geographical distribution of the Observational studies after 11th of March 2020.

To understand the monthly Research study completion rate as per geographic distribution of the Research.

Secondary Outcomes of the Study To understand the statistical correlation of the interventional studies Research with developed, developing and under developed countries.

To understand the statistical correlation of the observational studies Research with developed, developing and under developed countries.

To understand the statistical correlation of the Drug based interventional studies Research with developed, developing and under developed countries.

To understand the statistical correlation of the Diagnostic test based interventional studies Research with developed, developing and under developed countries.

To understand the statistical correlation of the Device based interventional studies Research with developed, developing and under developed countries.

Methodology WHO-compliant registries will be explored for completed COVID-19 Research articles.

Inclusion Criteria Interventional studies in the WHO-compliant registries database which are registered and completed after 11th of March 2020 until 15th of August 2020.

Observational studies in the WHO-compliant registries database which are registered and completed after 11th of March 2020 until 15th of August 2020.

Exclusion Criteria Interventional studies in the WHO-compliant registries database which are registered and completed before 11th March 2020.

Observational studies in the WHO-compliant registries database which are registered and completed before 11th March 2020.

The articles selected from the WHO-compliant registries database will be categorized as per following relevance:

Interventional Studies: Theses studies will be further categorized based on type of Intervention. Inteventional studies can be Drug, Diagnostic tests, Rehabilitation, Procedure, Device, Behavioral, Dietary supplement, Biological, Physiotherapy & Others types of Interventional study.

Observational Studies: Prospective and Retrospective Observational studies.

The Studies will be mapped according to the Country where the Research is completed and the type of Research.

Type of Variables studied in this Study 6 Continuous variables are studied in this Study Number of Interventional Studies (Continuous variable) Number of Observational Studies (Continuous variable) Number of Drug based Interventional Study (Continuous variable) Number of Diagnostic test based interventional study (Continuous variable) Number of Device based interventional study (Continuous variable) Monthly Research study completion rate (Continuous variable)

8 Categorical variables will be studies in this study Interventional Study (Categorical variable) Observational Study (Categorical variable) Developed country (Categorical variable) Developing country (Categorical variable) Under developed country (Categorical variable) Drug based Interventional Study (Categorical variable) Diagnostic test based interventional study (Categorical variable) Device based interventional study (Categorical variable)

Statistical Analysis Data analysis will be carried out using SPSS 22.00 (Stata Corp, College Station, TX, USA). The Data obtained will be analysed for the normal distribution. If the data follows normal distribution curve, Pearson Correlation statistical test will be used to assess the Correlation of categorical and continuous variables. If the data does not follow normal distribution curve, Spearman Correlation or Chi square statistical test will be used to assess the Correlation of Categorical and continuous variables. The p-value (significance level) of the correlation will be determined. If the p-value is <5%, then the correlation between variables analysed will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

Interventional studies in the WHO-compliant registries database which are registered and completed after 11th of March 2020 until 15th of August 2020.

Observational studies in the WHO-compliant registries database which are registered and completed after 11th of March 2020 until 15th of August 2020.

Exclusion Criteria:

Interventional studies in the WHO-compliant registries database which are registered and completed before 11th March 2020.

Observational studies in the WHO-compliant registries database which are registered and completed before 11th March 2020.

Min Age: 1 Year | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who are infected with COVID-19. Healthy Volunteers who respond to survey. Subjects who have recently recovered from COVID-19 infection.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-25 (Estimated); Primary Completion 2020-08-15 (Estimated); Study Completion 2020-09-20 (Estimated)

PRIMARY OUTCOMES:
Geographical distribution of the interventional studies after 11th of March 2020. | 15th of August 2020
  To understand the geographical distribution of the interventional studies after 11th of March 2020.
Geographical distribution of the Observational studies after 11th of March 2020. | 15th of August 2020
  To understand the geographical distribution of the Observational studies after 11th of March 2020.
Monthly Research study completion rate as per geographic distribution of the Research. | 15th of August 2020
  To understand the monthly Research study completion rate as per geographic distribution of the Research.

SECONDARY OUTCOMES:
Statistical correlation of the interventional studies Research with developed, developing and under developed countries. | 15th of August 2020
  To understand the statistical correlation of the interventional studies Research with developed, developing and under developed countries.
Statistical correlation of the observational studies Research with developed, developing and under developed countries. | 15th of August 2020
  To understand the statistical correlation of the observational studies Research with developed, developing and under developed countries.
Statistical correlation of the Drug based interventional studies Research with developed, developing and under developed countries. | 15th of August 2020
  To understand the statistical correlation of the Drug based interventional studies Research with developed, developing and under developed countries.
Statistical correlation of the Diagnostic test based interventional studies Research with developed, developing and under developed countries. | 15th of August 2020
  To understand the statistical correlation of the Diagnostic test based interventional studies Research with developed, developing and under developed countries.
Statistical correlation of the Device based interventional studies Research with developed, developing and under developed countries. | 15th of August 2020
  To understand the statistical correlation of the Device based interventional studies Research with developed, developing and under developed countries.

IPD SHARING:
Plan to Share IPD: No
The Research data will be extracted from the WHO-compliant registry databases.